CLINICAL TRIAL: NCT06130514
Title: The Comparison of Sympathetic Blockade of Stellate Ganglion Block and Thoracic Sympathetic Ganglion Block in Patients With Chronic Upper Extremity Neuropathic Pain: a Prospective Randomized and Comparative Clinical Trial
Brief Title: The Comparison of Sympathetic Blockade of Stellate Ganglion Block and Thoracic Sympathetic Ganglion Block
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University (Other)
Responsible Party: Principal Investigator, Jeeyoun Moon, Professor, Seoul National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2309-150-1472
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Chronic Pain; Neuropathic Pain; Complex Regional Pain Syndromes; Post Herpetic Neuralgia; Post Laminectomy Syndrome
MeSH Terms: conditions — Chronic Pain; Neuralgia; Complex Regional Pain Syndromes; Neuralgia, Postherpetic; post laminectomy syndrome | interventions — Ultrasonography; Fluoroscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided stellate ganglion block (US-guided SGB) (Active Comparator): In the case of ultrasound-guided stellate ganglion block, the patient is made to lie down and stellate ganglion block is performed by injecting 5 mL of 1% mepivacaine at the level of the 6th cervical vertebra using ultrasound.
  Interventions: Device: Ultrasound
- Fluoroscopy-guided thoracic sympathetic ganglion block (FS-guided TSGB) (Active Comparator): In the case of fluoroscopic device-guided thoracic sympathetic nerve block, place the patient prone and inject 3 mL of 1% mepivacaine at the level of the third thoracic vertebra to perform thoracic sympathetic nerve block.
  Interventions: Device: Fluoroscopy

INTERVENTIONS:
Device: Ultrasound — Ultrasound-guided stellate ganglion block with 1% mepivacaine 5 mL
  Arms: Ultrasound-guided stellate ganglion block (US-guided SGB)
Device: Fluoroscopy — Fluoroscopic-guided thoracic sympathetic ganglion block with 1% mepivacaine 3 mL
  Arms: Fluoroscopy-guided thoracic sympathetic ganglion block (FS-guided TSGB)

SUMMARY:
For patients scheduled to undergo upper limb sympathetic nerve block due to chronic neuropathic pain in the upper limb lasting more than 3 months, the ultrasound-guided stellate ganglion block group (S group) and the fluoroscopy-guided thoracic sympathetic nerve block group (T) Patients are randomly assigned 1:1 to one of the groups, and the procedure is performed. To evaluate the effectiveness of sympathetic nerve blockade, temperature changes in both palms are measured twice, 20 minutes before and 20 minutes after the procedure, using an infrared thermographer. Other variables related to the procedure are surveyed by outpatient visit or telephone before the procedure, after the procedure, before returning home, and 1 week and 1 month after the procedure.

DETAILED DESCRIPTION:
Patients aged 19 to 85 with upper limb pain are directly informed about the study, recruited, and enrolled at the Seoul National University Hospital Pain Center.

Before and after the procedure, continuous monitoring of electrocardiography, blood pressure, pulse rate, and oxygen saturation is carried out.

Before undergoing thoracic sympathetic ganglion block (TSGB) guided by fluoroscopy or ultrasound-guided stellate ganglion block (SGB), the temperature of both palms is measured using an infrared thermometer. Prior to the procedure, Doppler mode ultrasound equipment is used to measure blood flow velocity in the upper limb arteries (brachial artery).

In the case of ultrasound-guided stellate ganglion block, the patient is placed in a supine position, and the procedure is performed using ultrasound guidance to inject 5 mL of 1% mepivacaine at the level of C6. For fluoroscopy-guided thoracic sympathetic ganglion block, the patient is positioned prone, and 3 mL of 1% mepivacaine is injected at the level of T3. In both cases, the procedure is performed by a specialist with a rank of professor or higher who specializes in pain management.

After the procedure, the palm temperature is measured again 20 minutes later using an infrared thermometer.

Blood flow velocity in the upper limb arteries (brachial artery) is also measured 20 minutes post-procedure using Doppler mode ultrasound equipment.

Additionally, various procedure-related variables are assessed through outpatient visits or telephone surveys conducted before the procedure, at discharge, one week post-procedure, and four weeks post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with 19 - 85 years
* Patients with chronic upper extremity pain that lasts for more than 3 months
* Neuropathic pain conditions such as postherpetic neuralgia, complex regional pain syndrome, post laminectomy syndrome of cervical spine
* Patients judged to require sympathetic blockade by pain physician

Exclusion Criteria:

* Patient refusal
* Presence of upper limb vascular disorders
* History of previous thoracic sympathetic ganglion removal or neurolysis
* Abnormal findings in blood coagulation tests
* Systemic infection or local injection site infection
* Anatomical deformities at the injection site
* Allergic reactions to the injected medications
* Higher baseline hand temperature on the procedure side than the tympanic temperature (36.5°C) on pre-procedure thermography
* Other cases deemed inappropriate by the investigator

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2025-12-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
(1) Proportion of patients reaching > 1.5°C rise of temperature in the ipsilateral hand compared to the contralateral hand | 20 minutes after FS-guided thoracic sympathetic ganglion block or US-guided stellate ganglion block
  [ipsilateral hand temperature after the block - ipsilateral hand temperature before the block] - [contralateral hand temperature after the block - contralateral hand temperature before the block]

SECONDARY OUTCOMES:
(1) Difference of temperature change (°C) between ipsilateral hand and contralateral hand | 20 minutes after FS-guided thoracic sympathetic ganglion block or US-guided stellate ganglion block
  [ipsilateral hand temperature after the block - ipsilateral hand temperature before the block] - [contralateral hand temperature after the block - contralateral hand temperature before the block]
(2) Severity of pain | Time before block and 20 minutes and 1 week and 4weeks after FS-guided thoracic sympathetic ganglion block or US-guided stellate ganglion block
  11-point numerical rating scale (NRS)
(3) Patient satisfaction (PGIC scale) | 20 minutes and 1 week and 4 weeks after FS-guided thoracic sympathetic ganglion block or US-guided stellate ganglion block
  5-point Likert Scale
(4) Comparison of Korean version CISS(Cold Intolerance Symptom Severity) Questionnaire | Time before block and 4 weeks after FS-guided thoracic sympathetic ganglion block or US-guided stellate ganglion block
(5) Blood flow velocity measurement in upper extremity vessel(ipsilateral brachial artery) using ultrasound | Time before block and 20minutes after FS-guided thoracic sympathetic ganglion block or US-guided stellate ganglion block
  cm/s

CONTACTS AND LOCATIONS:
Overall Officials: Jee Youn Moon, MD, PhD, Principal Investigator — Seoul National University Hospital

REFERENCES:
- [Background] Kim YH, Kim SY, Lee YJ, Kim ED. A Prospective, Randomized Cross-Over Trial of T2 Paravertebral Block as a Sympathetic Block in Complex Regional Pain Syndrome. Pain Physician. 2019 Sep;22(5):E417-E424. PMID 31561653
- [Background] Kim J, Yun M, Han AH, Pauzi MF, Jeong JH, Yoo Y, Moon JY. Thoracic sympathetic ganglion blocks: real-world outcomes in 207 chronic pain patients. Reg Anesth Pain Med. 2024 Jul 8;49(7):528-535. doi: 10.1136/rapm-2023-104624. PMID 37726196
- [Background] Kim J, Lee HJ, Lee YJ, Lee CS, Yoo Y, Moon JY. Ultrasound-Guided Thoracic Paravertebral Block as a Sympathetic Blockade for Upper Extremity Neuropathic Pain: A Prospective Pilot Study. J Pain Res. 2020 Dec 14;13:3395-3403. doi: 10.2147/JPR.S285998. eCollection 2020. PMID 33363406
- [Background] Yoo HS, Nahm FS, Lee PB, Lee CJ. Early thoracic sympathetic block improves the treatment effect for upper extremity neuropathic pain. Anesth Analg. 2011 Sep;113(3):605-9. doi: 10.1213/ANE.0b013e3182274803. Epub 2011 Jul 21. PMID 21778335
- [Background] Day M. Sympathetic blocks: the evidence. Pain Pract. 2008 Mar-Apr;8(2):98-109. doi: 10.1111/j.1533-2500.2008.00177.x. PMID 18366465
- [Background] Rocha Rde O, Teixeira MJ, Yeng LT, Cantara MG, Faria VG, Liggieri V, Loduca A, Muller BM, Souza AC, de Andrade DC. Thoracic sympathetic block for the treatment of complex regional pain syndrome type I: a double-blind randomized controlled study. Pain. 2014 Nov;155(11):2274-81. doi: 10.1016/j.pain.2014.08.015. Epub 2014 Aug 19. PMID 25149143